CLINICAL TRIAL: NCT03928418
Title: Mobile Technology to Extend Clinic-based Counseling for HIV+s in Uganda
Acronym: EXTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Mbarara University of Science and Technology (Other); Syracuse University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA024990 (NIH); U01AA024990 (NIH)
Record Dates: First submitted 2019-04-10; First posted 2019-04-26 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use, Unspecified; HIV/AIDS
MeSH Terms: conditions — Alcohol Drinking; Acquired Immunodeficiency Syndrome | interventions — Technology; Spermine Synthase

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 3 arms. After the trial, participants in the standard of care arm, will be offered the intervention.
Who Masked: Investigator
Masking Description: The Research Assistant, who will collect study data including the study questionnaire and biological specimens for testing, will be blinded to the participants' study arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Phone Call Booster Arm (Experimental): The live phone call arm will include in-person counseling during 2 quarterly clinic visits plus live booster phone calls every three weeks in the interim.
  Interventions: Behavioral: In-person counseling session; Behavioral: Live phone call booster session
- Technology Booster Arm (Experimental): The technology booster arm will include in-person counseling during 2 quarterly clinic visits plus tech (choice of SMS or IVR) boosters once to twice weekly in the interim.
  Interventions: Behavioral: In-person counseling session; Behavioral: Technology (IVR or SMS) booster session
- Standard of Care (SOC) Arm (No Intervention): The standard of care (SOC) control (brief unstructured advice, with a wait-listed intervention).

INTERVENTIONS:
Behavioral: In-person counseling session — Brief alcohol reduction counseling is provided by a trained counselor to the study participant at the HIV clinic during two sessions that are 3 months apart.
  Arms: Live Phone Call Booster Arm; Technology Booster Arm
Behavioral: Live phone call booster session — Brief alcohol reduction counseling booster sessions every 3 weeks delivered via a live phone call from a trained counselor to the study participant given within 3 months and in between two in-person counseling sessions.
  Arms: Live Phone Call Booster Arm
Behavioral: Technology (IVR or SMS) booster session — Brief alcohol reduction counseling booster sessions once to twice a week delivered via a choice of interactive voice response (IVR) or short message service (SMS) phone technology to the study participant given within 3 months and in between two in-person counseling sessions.
  Arms: Technology Booster Arm

SUMMARY:
The EXTEND study is a randomized controlled trial to compare the uptake and acceptability, efficacy, and cost of methods of delivery of an alcohol intervention in reducing unhealthy alcohol use and increasing viral suppression among HIV positive persons in Uganda. The study arms are (a) in-person counseling during 2 quarterly clinic visits plus live booster phone calls every three weeks in the interim (b) in-person counseling during 2 quarterly clinic visits plus tech (choice of SMS or IVR) boosters once to twice weekly in the interim; and (c) standard of care (SOC) control (brief unstructured advice, with a wait-listed intervention).

DETAILED DESCRIPTION:
Alcohol consumption is a critical driver of HIV outcomes, especially in sub-Saharan Africa (SSA), where both are extremely common. Heavy alcohol use has been associated with reduced antiretroviral adherence, decreased HIV suppression, and increased mortality among those with HIV. Thus, reducing unhealthy alcohol use may improve HIV outcomes and is a high priority worldwide. Screening and brief counseling for alcohol use, especially multi-session approaches, have shown evidence for reducing alcohol use in resource rich settings and among persons with HIV. However, there are significant cost and human resource barriers to multiple session interventions in SSA, and it is not known whether alcohol interventions can improve HIV outcomes. Thus, the long-term goal of the EXTEND study is to develop and test interventions to reduce alcohol consumption and improve HIV outcomes, that can be feasibly integrated into routine HIV care in SSA.

Multi-session interventions that combine in-person visits with booster phone calls to reinforce the in-person counseling have shown good efficacy. Because cell phone use in Uganda is high, phone-based booster sessions conducted in-between the in-person sessions (that coincide with regularly scheduled clinic visits) may be feasible. However, phone-based booster sessions delivered by a live counselor ("live boosters") can be costly, time-consuming, limited to working hours, and dependent on good phone connections. Alternatively, automated cell phone-based booster sessions ("tech boosters"), can be conducted via interactive systems such as two-way Short Message Service (SMS, i.e. text messaging) or Interactive Voice Response (IVR) that allow for brief interactive sessions, with messages that are tailored to the participants' drinking goals and gender. Such automated tailored mobile phone-based interventions have been successful in improving several health behaviors in diverse populations. However, the uptake, acceptability, cost, and efficacy of live and tech booster calls for interventions for reducing alcohol use and improving HIV outcomes in SSA is not known. The investigators hypothesize that automated mobile phone-based technology can be leveraged as an efficacious way to implement multi-session alcohol interventions at a low burden and cost to both providers and patients in low resource settings.

Objectives

The EXTEND study is a randomized controlled trial (RCT) with a goal of estimating the uptake and acceptability, preliminary efficacy, and cost of methods of delivery of an intervention to reduce unhealthy drinking and HIV viral failure among persons in HIV care in rural Uganda (n=270). The RCT study arms are:

1. in-person counseling during 2 quarterly clinic visits plus live booster phone calls every three weeks in the interim;
2. in-person counseling during 2 quarterly clinic visits plus tech (choice of SMS or IVR) boosters once to twice weekly in the interim; and
3. standard of care (SOC) control (brief unstructured advice, with a wait-listed intervention).

This study will be conducted in a large rural Ugandan HIV clinic. The end products of this study will be the preliminary comparisons of key outcomes to estimate effect sizes and inform the design of a future large-scale trial. The long-term aim is to implement interventions that reduce alcohol use and improve HIV outcomes feasibly and at low cost in low resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older;
* HIV positive;
* On ART for at least six months;
* Reported alcohol use in the prior year at clinic entry;
* Fluency in Runyakole;
* Living within two hours travel time from the clinic;
* Owning or having daily access to a cell phone;
* Screening positive on the AUDIT-C

Exclusion Criteria:

* Plans to move out of the catchment area within 6 months;
* Unable to provide informed consent.
* Participation in another research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Hahn, PhD, MA, Principal Investigator — University of California, San Francisco
Locations (1):
- Mbarara University of Science and Technology/Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the final de-identified dataset from this study readily available for research purposes to other individuals in the scientific community. Data will be shared with the scientific community at large by posters and presentations at local, national, and international scientific meetings, as well as via peer- reviewed publications.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the RCT is concluded and data analyses are completed by the study team.
Access Criteria: The data and associated documentation will be made available to users only under a data-sharing agreement with the study investigators that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. User registration is required in order to access or download files. As part of the registration process, users must agree to the conditions of use governing access to the public release of data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource.

REFERENCES:
- [Background] Hahn JA, Woolf-King SE, Muyindike W. Adding fuel to the fire: alcohol's effect on the HIV epidemic in Sub-Saharan Africa. Curr HIV/AIDS Rep. 2011 Sep;8(3):172-80. doi: 10.1007/s11904-011-0088-2. PMID 21713433
- [Background] Hasin DS, Aharonovich E, O'Leary A, Greenstein E, Pavlicova M, Arunajadai S, Waxman R, Wainberg M, Helzer J, Johnston B. Reducing heavy drinking in HIV primary care: a randomized trial of brief intervention, with and without technological enhancement. Addiction. 2013 Jul;108(7):1230-40. doi: 10.1111/add.12127. Epub 2013 Apr 17. PMID 23432593
- [Background] Jonas DE, Garbutt JC, Amick HR, Brown JM, Brownley KA, Council CL, Viera AJ, Wilkins TM, Schwartz CJ, Richmond EM, Yeatts J, Evans TS, Wood SD, Harris RP. Behavioral counseling after screening for alcohol misuse in primary care: a systematic review and meta-analysis for the U.S. Preventive Services Task Force. Ann Intern Med. 2012 Nov 6;157(9):645-54. doi: 10.7326/0003-4819-157-9-201211060-00544. PMID 23007881
- [Background] Finitsis DJ, Pellowski JA, Johnson BT. Text message intervention designs to promote adherence to antiretroviral therapy (ART): a meta-analysis of randomized controlled trials. PLoS One. 2014 Feb 5;9(2):e88166. doi: 10.1371/journal.pone.0088166. eCollection 2014. PMID 24505411
- [Background] Crawford J, Larsen-Cooper E, Jezman Z, Cunningham SC, Bancroft E. SMS versus voice messaging to deliver MNCH communication in rural Malawi: assessment of delivery success and user experience. Glob Health Sci Pract. 2014 Jan 28;2(1):35-46. doi: 10.9745/GHSP-D-13-00155. eCollection 2014 Feb. PMID 25276561
- [Derived] Gichane MW, Camlin CS, Getahun M, Emenyonu N, Woolf-King S, Sanyu N, Katusiime A, Fatch R, Muyindike W, Hahn JA. Understanding Patients' Experiences with a Brief Alcohol Reduction Intervention among People Living with HIV in Uganda: A Qualitative Study. Subst Use Misuse. 2023;58(13):1714-1721. doi: 10.1080/10826084.2023.2244066. Epub 2023 Aug 8. PMID 37551890
- [Derived] Hahn JA, Fatch R, Emenyonu NI, Sanyu N, Katusiime A, Levine B, John Boscardin W, Chander G, Hutton H, Camlin CS, Woolf-King SE, Muyindike WR. Effect of two counseling interventions on self-reported alcohol consumption, alcohol biomarker phosphatidylethanol (PEth), and viral suppression among persons living with HIV (PWH) with unhealthy alcohol use in Uganda: A randomized controlled trial. Drug Alcohol Depend. 2023 Mar 1;244:109783. doi: 10.1016/j.drugalcdep.2023.109783. Epub 2023 Jan 21. PMID 36706675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment occurred from September 2019 through December 2020. 997 persons were screened; 272 unique individuals were enrolled and randomized. The first 3 people were enrolled as pilot participants and are excluded from all analyses, leaving 269 total persons for analysis.
Pre-assignment Details: The first 3 individuals enrolled in the study were considered "pilot" participants. They were randomized to one of the three study arms separately from the randomization for the main study participants. They are excluded from all analyses.
Period: Overall Study
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Started | 91 | 91 | 90
Pilot Participant (The first 3 participants enrolled in the study were pilot participants - they are included in the total number started, but were excluded from all analyses.) | 1 | 1 | 1
6-month Visit ((excluding pilot participants)) | 83 | 86 | 85
Completed ((excluding pilot participants)) | 85 | 87 | 84
Not Completed | 6 | 4 | 6
Not completed — Lost to Follow-up | 5 | 3 | 5
Not completed — Pilot participant - excluded from analyses | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: (1 person was found to have been enrolled in the SOC arm twice [protocol violation]; they are included only once.)
Groups:
- Total: Total of all reporting groups
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm | Total
Number analyzed (Participants) | 90 | 90 | 89 | 269
Age, Categorical [Count of Participants; unit: Participants] — Population: n=1 SOC participant missing age
  Participants
    number analyzed (Participants) | 90 | 90 | 88 | 268
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 89 | 90 | 85 | 264
    >=65 years | 1 | 0 | 3 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: n = 1 SOC participant missing age.
  years
    number analyzed (Participants) | 90 | 90 | 88 | 268
    (all) | 40.0 [34.0 to 47.0] | 39.5 [32.0 to 46.0] | 38.5 [33.0 to 46.0] | 39.5 [33.0 to 46.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 30 | 93
  Male | 57 | 60 | 59 | 176
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 90 | 90 | 89 | 269

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use Measured by Self Report
Description: Number of days drinking in the prior 21 days, as reported on the alcohol use timeline follow-back
Time Frame: At 6 and 9 month visits (3 and 6 months post intervention).
Population: The overall number of participants analyzed is the number of participants with self-reported alcohol use data at 6 months or 9 months.
Measure: Mean (95% Confidence Interval); unit: drinking days
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 85 | 87 | 85
drinking days
  At 6 month visit: number analyzed (Participants) | 83 | 86 | 85
  At 6 month visit | 2.9 [2.6 to 3.3] | 3.0 [2.6 to 3.4] | 5.5 [5.0 to 6.1]
  At 9 month visit: number analyzed (Participants) | 85 | 87 | 84
  At 9 month visit | 2.2 [1.9 to 2.5] | 2.8 [2.4 to 3.1] | 5.5 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Live Phone Call Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value comparing live call booster to SOC arm: p < 0.001 (calculated); Mixed effects model; random effects for participants; fixed effects for sex, baseline # of drinking days, visit, arm, interaction btwn visit and arm; Mean Difference (Net) = 3.5, 95% CI 2-sided [2.1 to 4.9] — SOC arm minus live call booster arm reported here
Statistical Analysis 2: Comparison: Technology Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value comparing technology booster to SOC arm: p < 0.001 (calculated); [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 3.6, 95% CI 2-sided [2.2 to 5.1] — SOC arm minus technology booster arm reported here

2. Primary Outcome: Change in Alcohol Use Measured by the Alcohol Biomarker, Phosphatidylethanol (PEth)
Description: Alcohol biomarker phosphatidylethanol (PEth) level will be used as an objective measure of prior 21-day alcohol use to confirm the findings obtained using self-report.
Time Frame: At 6 and 9 month visits (3 and 6 months post intervention).
Population: The overall number of participants analyzed is the number of participants with PEth alcohol biomarker data at 6 months or 9 months. n = 1 SOC participant was missing PEth from their 6 month visit.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 85 | 87 | 84
ng/mL
  At 6 month visit: number analyzed (Participants) | 83 | 86 | 84
  At 6 month visit | 376.9 [259.6 to 494.1] | 506.2 [386.1 to 626.3] | 396.9 [290.5 to 503.4]
  At 9 month visit | 313.8 [220.3 to 407.4] | 500.8 [340.2 to 661.3] | 396.2 [288.1 to 504.3]
Statistical Analysis 1: Comparison: Live Phone Call Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.643, Mixed Models Analysis — p-value comparing live call booster arm to SOC arm: p = 0.643; Mixed effects model; random effects for participants; fixed effects for sex, baseline PEth level, visit, arm, interaction btwn visit and arm; Mean Difference (Net) = 36.4, 95% CI 2-sided [-117.5 to 190.3] — SOC arm minus live call booster arm reported here
Statistical Analysis 2: Comparison: Technology Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.711, Mixed Models Analysis — p-value comparing technology booster arm to SOC arm: p = 0.711; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -30.9, 95% CI 2-sided [-194.8 to 132.9] — SOC arm minus technology booster arm reported here

3. Primary Outcome: Percentage of Participants With HIV Viral Suppression
Description: Undetectable HIV viral load measured through plasma HIV viral load measurements.
Time Frame: At 9 month visit (6 months post intervention).
Population: n = 5 participants in the live phone call booster arm and n = 3 participants in the technology booster arm were missing viral load results at their 9 month visits and are excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 80 | 84 | 84
percentage of participants | 95.0 [87.7 to 98.6] | 94.1 [86.7 to 98.0] | 92.9 [85.1 to 97.3]
Statistical Analysis 1: Comparison: Live Phone Call Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.515, Regression, Logistic — p-value comparing live call booster arm to SOC: p = 0.515; Mean Difference (Net) = -2.3, 95% CI 2-sided [-9.3 to 4.7] — SOC minus live call booster arm presented here
Statistical Analysis 2: Comparison: Technology Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.801, Regression, Logistic — p-value comparing technology booster arm to SOC: p = 0.801; Mean Difference (Net) = -0.9, 95% CI 2-sided [-8.3 to 6.4] — SOC minus technology booster arm presented here

4. Secondary Outcome: Percentage of Participants With Unhealthy Alcohol Use Via the AUDIT-C.
Description: Unhealthy alcohol use via the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), in the prior 3 months. The AUDIT-C ranges from 0-12. A score of 0 reflects no alcohol use; a score of 3 or higher in adult women or 4 or higher in men is considered positive for unhealthy alcohol use.
Time Frame: At 6 and 9 month visits (3 and 6 months post-intervention)
Population: Participants included are those with AUDIT-C data available at the 6- and 9-month visits.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 85 | 87 | 84
percentage of participants
  At 6 month visit: number analyzed (Participants) | 83 | 86 | 84
  At 6 month visit | 43.4 [32.5 to 54.7] | 46.5 [35.7 to 57.6] | 66.7 [55.5 to 76.6]
  At 9 month visit | 32.9 [23.1 to 44.0] | 40.2 [29.9 to 51.3] | 69.0 [58.0 to 78.7]
Statistical Analysis 1: Comparison: Live Phone Call Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value comparing live call booster arm to SOC: p < 0.001 (calculated); Mixed effects model; random effects for participants; fixed effects for sex, baseline alcohol use, visit, arm, interaction btwn visit and arm; Mean Difference (Net) = 28.9, 95% CI 2-sided [17.0 to 40.7] — SOC minus live call booster arm presented here
Statistical Analysis 2: Comparison: Technology Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value comparing technology booster arm to SOC: p < 0.001 (calculated); [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = 24.9, 95% CI 2-sided [13.0 to 36.8] — SOC minus technology booster arm presented here

5. Secondary Outcome: Number of Heavy Drinking Days in the Prior 21 Days
Description: The number of heavy drinking days in the prior 21 days will be defined as the number of days from the alcohol use timeline follow-back with ≥4/≥5 drinks reported by females/males, respectively, in the prior 21 days.
Time Frame: At 6 and 9 month visits (3 and 6 months post intervention).
Population: At 6 month visit: live call booster arm (n=83); technology booster arm (n=86); SOC arm (n=85).
  At 9 month visit: live call booster arm (n=85); technology booster arm (n=87); SOC arm (n=84).
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 85 | 87 | 85
days
  At 6 month visit: number analyzed (Participants) | 83 | 86 | 85
  At 6 month visit | 1.2 [1.0 to 1.5] | 1.4 [1.1 to 1.7] | 3.6 [3.2 to 4.0]
  At 9 month visit: number analyzed (Participants) | 85 | 87 | 84
  At 9 month visit | 0.6 [0.5 to 0.8] | 1.5 [1.3 to 1.8] | 3.3 [2.9 to 3.7]
Statistical Analysis 1: Comparison: Live Phone Call Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value comparing live call booster arm to SOC: p = 0.002; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = 4.4, 95% CI 2-sided [1.6 to 7.3] — SOC arm minus live call booster arm presented here
Statistical Analysis 2: Comparison: Technology Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value comparing technology booster arm to SOC: p = 0.003; [statistical method as in outcome 4, analysis 1]; Mean Difference (Net) = 4.3, 95% CI 2-sided [1.5 to 7.2] — SOC arm minus technology booster arm presented here

6. Secondary Outcome: Cluster of Differentiation-4 (CD4) Cell Count
Description: CD4 cell count of participants measured through plasma CD4 measurements.
Time Frame: At nine months (6 months post intervention).
Population: CD4 count data were not collected and as such, this analysis was not completed. We had intended to extract CD4 cell counts from HIV clinic records; however, the clinic discontinued CD4 testing when viral load monitoring became routine.
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percent of Antiretroviral Therapy (ART) Adherence in the Prior 30 Days.
Description: Percent self-reported antiretroviral therapy (ART) adherence in the prior 30 days. This measure was defined as the lower of two self-reported measures of ART adherence in the prior 30 days: 1. a visual analog scale: a line ranging from 0% (no doses) to 100% (all doses) on which participants indicated how many of their ART doses they had taken, and 2. the percentage of days that the participant reported taking all of their ART pills.
Time Frame: At 6 and 9 month visits (3 and 6 months post intervention).
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: adherence percentage
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 85 | 87 | 85
adherence percentage
  At 6 month visit: number analyzed (Participants) | 83 | 86 | 85
  At 6 month visit | 92.3 [89.4 to 95.2] | 91.6 [88.4 to 94.7] | 90.4 [88.2 to 92.7]
  At 9 month visit: number analyzed (Participants) | 85 | 87 | 84
  At 9 month visit | 93.3 [91.3 to 95.4] | 93.3 [90.3 to 96.2] | 92.8 [91.0 to 94.5]
Statistical Analysis 1: Comparison: Live Phone Call Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.610, Mixed Models Analysis — p-value comparing live call booster arm to SOC arm: p = 0.610; Mixed effects model; random effects for participants; fixed effects for sex, baseline ART adherence, visit, arm, interaction btwn visit and arm; Mean Difference (Net) = -0.8, 95% CI 2-sided [-3.8 to 2.2] — SOC minus live call booster arm presented here
Statistical Analysis 2: Comparison: Technology Booster Arm vs Standard of Care (SOC) Arm; Test type: Superiority; p = 0.474, Mixed Models Analysis — p-value comparing technology booster arm to SOC arm: p = 0.474; [statistical method as in outcome 7, analysis 1]; Mean Difference (Net) = -1.1, 95% CI 2-sided [-4.1 to 1.9] — SOC minus technology booster arm presented here

8. Secondary Outcome: Booster Uptake - Completion
Description: Technology booster uptake is defined as the percentage of technology booster sessions initiated by the system, in which the participant answered all the required questions.
  Live booster call uptake is defined as the percentage of live booster calls attempted, that were completed by the participant.
  This was a descriptive analysis of the mean percentage of boosters completed per participant.
Time Frame: 3 months
Population: 0 participants from the SOC arm are included here because they did not receive boosters.
Measure: Mean (95% Confidence Interval); unit: % boosters completed
Units Other Than Participants: Boosters attempted
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 90 | 90 | 0
Number analyzed (Boosters attempted) | 290 | 2114 | 0
% boosters completed | 86.5 [81.8 to 91.3] | 44.7 [33.4 to 51.1] |

9. Secondary Outcome: Booster Uptake - Counselor Call-back Requests
Description: Number of participants in the technology booster arm who requested at least one counselor call-back during their technology session.
Time Frame: 3 months
Population: This descriptive analysis was only completed among participants in the technology booster arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 0 | 90 | 0
Participants |  | 57 |

10. Secondary Outcome: Booster Satisfaction - Client Satisfaction Scale-8
Description: Intervention satisfaction in each arm will be assessed using the Client Satisfaction Scale-8 (CSQ-8). The CSQ-8 is an 8-item questionnaire used to assess satisfaction with services in health and human services. The response options (1. Quite dissatisfied, 2. Indifferent or mildly dissatisfied, 3. Mostly satisfied, 4. Very satisfied) range from very negative to very positive, correlating with low to high satisfaction. The scale ranges from 25-100, with higher numbers indicating higher satisfaction.
Time Frame: At 6 month visit (3 months post intervention)
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 83 | 86 | 85
score on scale | 93.3 [91.9 to 94.8] | 93.1 [91.8 to 94.5] | 90.0 [88.2 to 91.8]

11. Secondary Outcome: Booster Satisfaction - Usability
Description: Usability was assessed in the technology booster arm via the System Usability Scale (SUS), used to evaluate new technology, and the proportions that chose short message service (SMS, text message) over interactive voice recognition (IVR) as the mode of booster delivery, overall and by reading literacy (yes/no). The System Usability Scale is a 10-item questionnaire; raw score totals range from 0 to 40 with higher scores indicating better usability.
Time Frame: At 6 month visit (3 months post intervention).
Population: System usability was assessed only within the technology booster arm.
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
Number analyzed (Participants) | 0 | 86 | 0
score on scale |  | 34.9 [34.2 to 35.5] |

12. Secondary Outcome: IVR Chosen as Technology Booster Mode
Description: Participants in the technology booster arm chose to receive the boosters via either interactive voice response (IVR) or short message service (SMS, text). We report here on the number of participants choosing IVR among technology booster arm participants overall, and by literacy status.
Time Frame: 3 months
Population: Participants randomized to the technology booster arm, included in this descriptive analysis overall and stratified by literacy status.
Measure: Count of Participants; unit: Participants
Groups:
- Technology Booster Arm - All Participants: The technology booster arm will include in-person counseling during 2 quarterly clinic visits plus tech (choice of SMS or IVR) boosters once to twice weekly in the interim.
  In-person counseling session: Brief alcohol reduction counseling is provided by a trained counselor to the study participant at the HIV clinic during two sessions that are 3 months apart.
  Technology (IVR or SMS) booster session: Brief alcohol reduction counseling booster sessions once to twice a week delivered via a choice of interactive voice response (IVR) or short message service (SMS) phone technology to the study participant given within 3 months and in between two in-person counseling sessions.
- Technology Booster Arm - Literate Participants: Participants in the technology booster arm, who were literate/somewhat literate.
- Technology Booster Arm - Not Literate Participants: Participants in the technology booster arm, who were not literate.
Arm/Group | Technology Booster Arm - All Participants | Technology Booster Arm - Literate Participants | Technology Booster Arm - Not Literate Participants
Number analyzed (Participants) | 90 | 77 | 13
Participants | 59 | 46 | 13

13. Other Pre Specified Outcome: Cost Methodology
Description: To determine costs, the investigators collected data to capture all relevant direct (e.g. equipment) and indirect (e.g. administrative), fixed (or 'start-up') and variable (or 'recurring') costs related to the intervention activities. Costs were differentiated by intervention component (e.g. clinic-based counseling versus remote booster sessions) and by booster session mode of delivery (i.e. live booster versus tech booster, and between SMS and IVR tech boosters). Total observed costs (US$) were collected by booster session delivery mode and divided by the number of participants who received that booster session type. That includes participants who were randomized to each arm as well as participants randomized to the standard of care (SOC) arm who received the intervention after a wait-list control period. No individual-level data were collected; because of this, no measures of dispersion exist.
Time Frame: Live Phone Call and Technology Booster Arms: from baseline to 3 months; for SOC wait-listed participants: from 9 months to 12 months.
Population: The costing analysis was conducted for the study intervention booster session mode of delivery (ie. live call, interactive voice recognition (IVR) and short message service (SMS) technology boosters). Participants from the SOC arm who received the intervention after a wait-list control period are also included here.
Measure: Number; unit: cost (US$) per participant
Groups:
- Technology Booster Arm - SMS: The technology booster arm will include in-person counseling during 2 quarterly clinic visits plus boosters once to twice weekly in the interim. This group was randomized to the technology booster arm, and chose SMS as the mode of booster delivery.
  In-person counseling session: Brief alcohol reduction counseling is provided by a trained counselor to the study participant at the HIV clinic during two sessions that are 3 months apart.
  Technology (SMS) booster session: Brief alcohol reduction counseling booster sessions once to twice a week delivered via short message service (SMS) phone technology to the study participant given within 3 months and in between two in-person counseling sessions.
- Technology Booster Arm - IVR: The technology booster arm will include in-person counseling during 2 quarterly clinic visits plus boosters once to twice weekly in the interim. This group was randomized to the technology booster arm, and chose IVR as the mode of booster delivery.
  In-person counseling session: Brief alcohol reduction counseling is provided by a trained counselor to the study participant at the HIV clinic during two sessions that are 3 months apart.
  IVR booster session: Brief alcohol reduction counseling booster sessions once to twice a week delivered via interactive voice response (IVR) phone technology to the study participant given within 3 months and in between two in-person counseling sessions.
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm - SMS | Technology Booster Arm - IVR
Number analyzed (Participants) | 160 | 40 | 61
cost (US$) per participant | 144.27 | 312.79 | 315.45

ADVERSE EVENTS:
Time Frame: 9 months
Description: The definition of adverse event and/or serious adverse event did not differ from the clinicaltrials.gov definitions.
  Adverse events were recorded during routine study visits when self reported by participants.
Arm/Group | Live Phone Call Booster Arm | Technology Booster Arm | Standard of Care (SOC) Arm
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/90 | 0/90 | 0/89
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Live Phone Call Booster Arm (N=90) | Technology Booster Arm (N=90) | Standard of Care (SOC) Arm (N=89)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study of the impact of the interventions on HIV viral suppression was limited, as non-suppression is low in Uganda and was not an eligibility criterion. Ability to prevent cross-contamination across study arms was limited but we felt the likelihood of this was low as the intervention occurred at a large clinic. Persons with severe alcohol use disorder were not excluded, potentially limiting findings. The single site and occurrence of a global pandemic limit the generalizability of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03928418/Prot_SAP_ICF_001.pdf